CLINICAL TRIAL: NCT00777855
Title: The Effects of Rifampin on the Pharmacokinetics of Warfarin in Healthy Volunteers.
Brief Title: Drug Interaction Study of Rifampin and Warfarin in Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: warfarin-6006
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: warfarin; pharmacokinetics; drug transporter; healthy volunteer; drug interaction; rifampin
MeSH Terms: interventions — Warfarin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- warfarin then warfarin plus rifampin (Experimental)
  Interventions: Drug: warfarin plus rifampin; Drug: warfarin

INTERVENTIONS:
Drug: warfarin plus rifampin — warfarin 7.5mg po x 1; rifampin 600mg IV x 1
Drug: warfarin — warfarin 7.5mg po x 1

SUMMARY:
The purpose of this study is to determine the importance of uptake drug transporters in the drug disposition of warfarin. We predict that the elimination of warfarin will be decreased when co-dosed with an inhibitor of uptake drug transporters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-60 years of age;
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam and laboratory evaluations;
* BMI between 18.5 - 30 kg/m2;
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or over-the-counter (OTC) medications (except acetaminophen);
* Subjects able to maintain adequate birth control during the study independent of hormonal contraceptive use;
* Be able to provide written informed consent and comply with requirements of the study;
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until completion of the entire study;
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 6pm the night before a study day until completion of that study day;
* Avoidance of contact sports and/or other activities with significant risk of trauma injury for 7 days after each study day.
* Fast from food and beverages at least 8 hours prior to medication dosing;
* Be able to read, speak and understand English

Exclusion Criteria:

* Subjects on prescription or chronic over-the counter medications (including hormonal contraceptives);
* Subjects with known allergy to warfarin and/or rifampin;
* Subjects who are not homozygous for cytochrome P450 2C9 (CYP2C9 *1) (known poor metabolizers).
* Subjects with a history or diagnosis of hemorrhagic tendencies or blood dyscrasias;
* Subjects with liver failure or liver function test (LFT) results >2x upper limit of normal;
* Subjects with clinically significant elevations in international normalized ratio (INR), prothrombin (PT), prothrombin time (PTT), serum creatinine (SCr), blood urea nitrogen (BUN) or other screening laboratory tests as determined by study physician;
* Subjects with Hct <30 mg/dL;
* Subjects with history of GI bleed or peptic ulcer disease;
* Subjects with a recent history of trauma;
* Subjects with a recent history of or upcoming plan of surgery;
* Subjects who smoke tobacco;
* Subjects with ongoing alcohol or illegal drug use;
* Subjects who are pregnant, lactating or attempting to conceive;
* Subjects unable to maintain adequate birth control during the study;
* Subjects unable to follow protocol instructions or protocol criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy non-smoking volunteers from community
Pre-assignment Details: All participants were medication free throughout study enrollment
Groups:
- Warfarin First, Then Warfarin+Rifampin: In a randomized, single-dose, two-period, crossover design, 5 participants received warfarin alone 7.5mg po; after a minimum of 14 days, participants received a 30-minute IV infusion of 600mg rifampin immediately followed by warfarin 7.5mg po.
- Warfarin+Rifampin First, Then Warfarin Alone: In a randomized, single-dose, two-period, crossover design, 5 participants received a 30-minute IV infusion of 600mg rifampin immediately followed by warfarin 7.5mg po; after a minimum of 14 days, participants received warfarin alone 7.5mg po.
Period: First Intervention
Arm/Group | Warfarin First, Then Warfarin+Rifampin | Warfarin+Rifampin First, Then Warfarin Alone
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout Period (>= 14 Days)
Arm/Group | Warfarin First, Then Warfarin+Rifampin | Warfarin+Rifampin First, Then Warfarin Alone
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Warfarin First, Then Warfarin+Rifampin | Warfarin+Rifampin First, Then Warfarin Alone
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive warfarin alone then warfarin+rifampin, and those randomized to receive warfarin+rifampin then warfarin alone in the crossover design
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: S- and R- Enantiomers of Warfarin (S-warfarin and R-warfarin) Area Under the Plasma Concentration-time Curve (AUC) From 0 to 12 Hours.
Description: Uptake effects on warfarin pharmacokinetics during time period of hepatic organic anion-transporting polypeptide (OATP) inhibition by rifampin. Blood collection 1, 2, 4, 6, 8, and 12 hours after warfarin dosing.
Time Frame: 0-12 hours after warfarin dosing
Population: Each of 10 participants received both treatments separated by a minimum of 14 days; treatment sequence was randomly assigned
Measure: Mean (Standard Deviation); unit: ng/ml*h
Groups:
- Warfarin: warfarin : warfarin 7.5mg po x 1
- Warfarin Plus Rifampin: warfarin plus rifampin : warfarin 7.5mg po x 1 immediately following rifampin 600mg IV x 1
Arm/Group | Warfarin | Warfarin Plus Rifampin
Number analyzed (Participants) | 10 | 10
ng/ml*h
  AUC (0-12 hours) of S-warfarin | 2,250 (340) | 2,230 (460)
  AUC (0-12 hours) of R-warfarin | 2,850 (460) | 2,930 (510)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity of S-warfarin and R-warfarin
Description: Analysis of all concentration-time data. Blood collection 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after warfarin dosing.
Time Frame: 0-120 hours after warfarin dosing
Population: Each of 10 participants received both treatments, in randomly assigned order, separated by a minimum of 14 days
Measure: Mean (Standard Deviation); unit: ng/ml*h
Arm/Group | Warfarin | Warfarin Plus Rifampin
Number analyzed (Participants) | 10 | 10
ng/ml*h
  AUC(0-infinity) of S-warfarin | 8,420 (1,090) | 7,410 (2,500)
  AUC(0-infinity) of R-warfarin | 18,600 (3,400) | 14,100 (4,100)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of S-warfarin and R-warfarin
Description: Blood collection 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after warfarin dosing.
Time Frame: 0-120 hours after warfarin dosing
Population: Each of 10 participants received both treatments, in randomly assigned order, separated by a minimum of 14 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Warfarin | Warfarin Plus Rifampin
Number analyzed (Participants) | 10 | 10
ng/ml
  Cmax of S-warfarin | 329 (70) | 303 (82)
  Cmax of R-warfarin | 375 (116) | 351 (85)

ADVERSE EVENTS:
Time Frame: 120 hours after warfarin dosing
Description: Each of 10 participants received 2 treatments (warfarin, with or without rifampin), in randomly assigned order, separated by a minimum of 14 days. Participants presented for venous blood collection and were assessed for adverse events at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after warfarin dosing.
Groups:
- Entire Study Population: Each of 10 participants received both study treatments, in randomly assigned sequence, separated by a minimum of 14 days
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes